CLINICAL TRIAL: NCT01232959
Title: Feasibility of Transvaginal Cholecystectomy
Acronym: TVC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Subjects not interested
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Juliane Bingener-Casey, PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-001167
Record Dates: First submitted 2010-10-28; First posted 2010-11-02 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Gallstones
Keywords: Gallbladder removal
MeSH Terms: conditions — Gallstones | interventions — Cholecystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transvaginal Surgery (Experimental): Gallbladder will be removed through the vagina
  Interventions: Device: Transvaginal Cholecystectomy

INTERVENTIONS:
Device: Transvaginal Cholecystectomy — A small incision is made in the vagina. An endoscope (flexible lighted camera tube) is inserted into the abdomen. An endoscope is normally used to examine your stomach or colon. A very small camera is placed in your abdomen at the belly button (5 mm, ¼ inch). This helps the surgeons to remove your gallbladder through the vagina. The procedure to separate your gallbladder from your body will be assisted by instruments placed through your abdomen and instruments placed in your vagina. The surgeon will remove the gallbladder by passing it though your vagina.
  Other Names: gallbladder removal

SUMMARY:
Today there are three different ways to remove a gallbladder with gallstones. Surgeons can remove the gallbladder through small incisions in the abdomen. This is called laparoscopic cholecystectomy. It is the current standard. It has replaced traditional open gallbladder surgery. Open gallbladder surgery is done with a large incision. A new way of removing the gallbladder in women is through the vagina. This is called transvaginal cholecystectomy. This study is being done to see if removing the gallbladder through the vagina will work for patients at Mayo Clinic Rochester. This is the first step of this research to test the procedure. In the future, other studies will examine the potential for less scarring and reduced pain. In this study the investigators will still make small incisions in the abdomen, they will be smaller than the standard procedure but you will still have some scars on your abdomen.

Some very early research reports say that some patients may have less pain with the transvaginal approach; however, the investigators do not know if the transvaginal route will have any effect on your overall health and quality of life.

This study will evaluate:

* Effectiveness of the surgery: ability to remove the gallbladder safely
* Effect of the operation on your body: change in pulse and blood pressure during the surgery, level of inflammation markers in your blood before and after the surgery
* Recovery from surgery in the hospital: how much pain you have, how much pain medication you need, how long you need to stay in the hospital, or nature of any surgical complications (problems)
* Overall recovery from surgery: general quality of life, abdominal symptoms

What is the new type of surgery?

The new type of surgery is called transvaginal cholecystectomy:

A small incision is made in the vagina. An endoscope (flexible lighted camera tube) is inserted into the abdomen. An endoscope is normally used to examine your stomach or colon. A very small camera is placed in your abdomen at the belly button (5 mm, ¼ inch). This helps the surgeons to remove your gallbladder through the vagina. The procedure to separate your gallbladder from your body will be assisted by instruments placed through your abdomen and instruments placed in your vagina. The surgeon will remove the gallbladder by passing it though your vagina.

DETAILED DESCRIPTION:
As technologic innovations in medicine continue to advance, less intrusive operative procedures are being developed. Natural Orifice Transluminal Endoscopic Surgery (NOTES) may represent a less invasive approach to the abdominal cavity. The access to the abdominal cavity through natural orifices such as the vagina has the benefit of decreased somato-sensory innervation. This venue might confer less pain and operative stress to the patient. The transvaginal approach has been suggested as a new surgical approach to gallbladder surgery (cholecystectomy). Approximately 700 transvaginal cholecystectomy procedures have been performed in medical centers around the world so far. Anecdotal data suggest that the patients experience less pain postoperatively and half of them may not require any pain medication. Currently, introduction of this new operative approach outside of a research study is not supported by national nor international societies.

We wish to demonstrate that the transvaginal approach is feasible for 10 patients with gallstone disease at Mayo Clinic Rochester (MCR).

Methods: Female patients seen by consultants from the Division of General and Gastrointestinal Surgery, who have an appropriate indication for elective cholecystectomy, will be offered a cholecystectomy via the transvaginal approach. After patient enrollment, baseline demographics, questionnaires and blood draws will be obtained. The patient will undergo a laparoscopic assisted transvaginal cholecystectomy by a dedicated surgical team, consisting of a gynecologist, a minimally invasive surgeon and a gastroenterologist. This approach will utilize a 5-mm umbilical trocar and a posterior colpotomy. Standard laparoscopic and flexible endoscopic instrumentation will be utilized along with recently introduced long flexible-tip laparoscopic instrumentation to remove the gallbladder. Intraoperative parameters will be recorded. Postoperatively blood draws and questionnaires will be repeated at specific intervals.

Data analysis will be mainly descriptive for this feasibility study. The collected material will serve as pilot data for a future comparative study of transvaginal cholecystectomy with standard laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion criteria

* Female patients undergoing elective cholecystectomy for cholelithiasis.

Exclusion criteria

* Male patients, patients <18 years or >65 years of age
* Pregnant patients
* Patients with prior pelvic surgery
* Patients with prior hepatobiliary surgery or other major abdominal surgery
* Patients with ASA class >3
* Patients with BMI >35
* Patients with risk factors for requiring an open cholecystectomy (e.g. possible gallbladder cancer, acute cholecystitis, jaundice)
* Patients who cannot provide consent for the study
* Patients not willing to participate in the study.
* Patients with common bile duct stones
* Patients with evidence of abdominal abscess or mass
* Patients with diffuse peritonitis
* Patients with a clinical diagnosis of sepsis
* Patients with coagulopathy or using anticoagulants or anti-platelet agents (aspirin up to 81mg/day acceptable)
* Patients with planned concurrent procedures
* Patients with a prior diagnosis of intra-abdominal adhesions
* Patients who are participating in any other investigational device or drug trial that has not yet completed the primary endpoint
* Patients with an enlarged uterus

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Feasibility measured by successful transvaginal removal of gallbladder | 1 year
  The procedure will be considered technically successful if at completion the cystic duct and artery have been clipped securely and the gallbladder has been removed through the transvaginal port. At the time of surgery, the procedure will be supervised with a laparoscope at all critical points. Conversion to a laparoscopic or open procedure is considered an incomplete transvaginal procedure.

SECONDARY OUTCOMES:
Safety and tolerability measured by individual and overall Adverse Events | Following each surgery but overall at 1 year
  1. Procedural complications recorded during transvaginal cholecystectomy.
  2. Complications resulting from endoscopic transvaginal cholecystectomy recorded at the time of surgery.
  3. Patients' post-operative clinical course for duration of three months, including routine follow up at about one week after the operation, vaginal exam after six weeks and follow-up with quality of life questionnaire at three months.
Pain Scores as measured on the Visual Analog Scale | 1 year
  One of the main endpoints of the study will be postoperative pain as measured by the visual analog scale. The scale will be measured in triplicate fashion. In addition to the visual analog scale, the amount and class of pain medication used will be collected.
Quality of Life measured through validated questionnaires | 1 year
  Data for the SF-12 and ASIS will be scaled and evaluated for correlation at baseline and postoperative day 7 with the Pearson coefficient. Change from baseline for each instrument will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Juliane Bingener-Casey, MD, Principal Investigator — Mayo Clinic